CLINICAL TRIAL: NCT07115875
Title: Improving Rates of Diagnostic Colonoscopy in Native Americans Through a Culturally Sensitive Digital Outreach Intervention
Brief Title: Improving Rates of Diagnostic Colonoscopy in Native Americans
Acronym: YVONNE-DX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 16811
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: CRC Screening; CRC (Colorectal Cancer)
Keywords: Mobile Health Technology; Telehealth; Digital Outreach
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The two factors (Outreach Type and Consultation Type) will be crossed with one another to create a total of four experimental conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Outreach and Telehealth Consultation (Experimental): The investigators will disseminate mHealth Outreach, using SMS texts with culturally relevant language and short videos that include personal narratives of patients and high-status Tribal members, to increase motivation to a schedule a diagnostic colonoscopy.
  Second, the investigators will try and overcome one refractory structural barrier to completing a diagnostic colonoscopy among Cheyenne and Arapaho Tribal members through telehealth. Cheyenne and Arapaho patients are required to visit the colonoscopy clinical facilities for both a pre-procedure appointment and the actual procedure. This process requires two round trips to a colonoscopy facility located in Lawton, OK, which is over 90 miles from the Clinton Indian Health Center. As a result, the investigators have proposed to test whether offering the pre-procedure as a telehealth consultation will overcome this transportation barriers.
  Interventions: Other: Digital Outreach
- In Person Consultation (Active Comparator): Participants randomized to In-Person Consultation will receive standard of care at IHS Lawton Hospital. Consultation includes a colonoscopy risk assessment (i.e., current medication use, risk of perforation and bleeding, ability to complete bowel prep).
  Interventions: Other: In Person consultation

INTERVENTIONS:
Other: Digital Outreach — Digital outreach interventions through focus groups. The study is based on narrative interventions that highlights culturally sensitive and values among Native American communities.
  Arms: mHealth Outreach and Telehealth Consultation
Other: In Person consultation — In-Person Consultation will receive standard of care at IHS Lawton Hospital. Consultation includes a colonoscopy risk assessment (i.e., current medication use, risk of perforation and bleeding, ability to complete bowel prep).
  Arms: In Person Consultation

SUMMARY:
Colorectal cancer (CRC) is the second-leading cause of cancer death in both men and women in the United States. Compared to national averages, Native Americans (NA) endure a disproportionate burden of CRC incidence and CRC-specific mortality. The long-term goal of this collaboration is to enhance health equity through the reduction of CRC disparities in morbidity, mortality, stage-at-diagnosis, and survival among NA. To do so, the primary focus of these efforts has been to improve processes that increase uptake of home stool screening. The overall objective is to leverage these relationships and infrastructure to now focus on improving rates of timely diagnostic colonoscopy follow up after an abnormal home stool screening.

DETAILED DESCRIPTION:
PURPOSE AND/OR HYPOTHESIS:

The proposed study is segmented into two study Stages. Stage 1 incorporates Study Aim 1, which will use focus groups to co-develop a digital outreach intervention with Native Americans. Focus groups will help better understand how the investigators can support timely screening for colorectal cancer in this community. This IRB submission is seeking OUHSC IRB approval to conduct Stage 1. Before conducting any data collection, the investigators will seek IHS Tribal IRB approval. Once approval has been received from both OUHSC and IHS IRB, analysis of the data collected from Stage 1 will then be used to inform Stage 2. To ensure NIH funding of this grant, OUHSC IRB approval must be achieved by November 30, 2025.

Stage 2 incorporates Study Aims 2 and 3. For those aims, the investigators will test the reach, feasibility, and potential efficacy of digital outreach intervention strategies (Aim 2) and the penetration, acceptability, and scalability of the digital outreach intervention strategies (Aim 3). Dr. Neil will submit an IRB modification to both OUHSC and IHS IRBs after data analysis from Stage 1 has been completed and prior to conducting any human subjects research in Stage 2.

Native Americans (NA) endure a disproportionate burden of colorectal cancer (CRC) incidence and CRC-specific mortality. Screening is an effective early detection strategy to decrease preventable CRC-related deaths, but NA have some of the lowest CRC screening rates. In Oklahoma, only 51% of NA are up to date with screening compared to nearly two-thirds of eligible US adults. Efforts to reduce disparities in screening rates have focused on increasing access to home stool screening. However, approximately one-half of NA in Oklahoma with an abnormal home stool test do not complete a required follow-up diagnostic colonoscopy. As time to colonoscopy after an abnormal home stool test is associated with greater diagnosis of late-stage disease and CRC mortality, innovative strategies are needed to increase rates of timely diagnostic colonoscopy follow up among NA in Oklahoma. The proposed study leverages an existing relationship with the Cheyenne and Arapaho Tribes to co-develop and pilot test two digital outreach interventions to increase rates of diagnostic colonoscopy. First, mobile health outreach (mHealth; SMS text and video messages) will attempt to increase motivation to schedule a diagnostic colonoscopy. In addition to receiving informational texts about how and why to schedule a colonoscopy, participants will also receive culturally sensitive videos that use personal narratives from NA patients and other high-status Cheyenne and Arapaho Tribal members (e.g., elders). Second, current clinic workflow requires Cheyenne and Arapaho patients to visit the colonoscopy clinical facilities for both a pre-visit appointment and the actual procedure. This process requires a minimum of two round trips to a colonoscopy facility of over 90 miles for most patients. The investigators will test whether a pre-visit telehealth consultation reduces transportation barriers. Our overarching hypothesis is that culturally sensitive digital outreach intervention will increase motivation, reduce structural barriers, and, thus, improve rates of diagnostic colonoscopy.

The first study aim will co-develop culturally sensitive digital outreach intervention strategies, guided by four focus groups of NA patients (6 participants per group, with a total of 24 participants) and a community advisory board.

The second study aim will determine reach, feasibility, and potential efficacy of intervention strategies testing an mHealth outreach vs. informational pamphlet and a telehealth vs. in-person pre-visit colonoscopy consultation among 140 NA patients. The primary outcome is potential efficacy, measured as rates of diagnostic colonoscopy 60 days post-randomization. The third aim will explore penetration, acceptability, and scalability of digital outreach intervention strategies. If effective, this first-of-its-kind and highly scalable approach offers a substantial public health impact to reduce avoidable CRC morbidity and mortality among NA patients by increasing rates of diagnostic colonoscopy.

EXPERIMENTAL DESIGN:

For Stage 1, there is no experimental design.

For Stage 2, Aim 2 will use a 2 x 2 factorial design: (Outreach Type, Factor 1) mHealth outreach vs. informational pamphlet; (Consultation Type, Factor 2) telehealth vs. in-person pre-visit colonoscopy consultation. The primary outcome is potential efficacy, measured as rates of diagnostic colonoscopy 60 days post-randomization. The third aim will explore penetration, acceptability, and scalability of digital outreach intervention strategies.

PROPOSED PROCEDURE:

For Stage 1, Aim 1, the proposed procedure is broken into three Phases. Phase 1 will co-develop the mHealth Outreach (i.e., SMS texts and videos) content in 4 focus groups (n=6-8 per group) of NA from in Oklahoma that from IHS Clinton Service Unit. Groups will be stratified by history of diagnostic colonoscopy (yes/no). Phase 2 will create the mHealth outreach message library. Phase 3 will employ a community advisory board (CAB) to discuss how best to integrate mHealth and Telehealth interventions into clinic workflows.

IMPORTANCE OF KNOWLEDGE REASONABLY EXPECTED TO RESULT FROM THE RESEARCH:

The long-term goal of this collaboration is to enhance health equity through the reduction of CRC disparities in morbidity, mortality, stage-at-diagnosis, and survival among NA. To do so, the primary focus of these efforts has been to improve processes that increase uptake of colorectal cancer screening and improve rates of timely diagnostic colonoscopy follow up after an abnormal home stool screening.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Live in Oklahoma
* Fluent in English
* Have access to email
* Identify as Native American or have a Certificate of Degree of Indian Blood

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Focus Group Strategy | 6 months
  The investigators will use focus groups to co-develop a digital outreach intervention with Native Americans. Focus groups will help better understand how the investigators can support timely screening for colorectal cancer in this community

SECONDARY OUTCOMES:
Digital Outreach Intervention Strategies | 6 months
  We will test the reach, feasibility, and potential efficacy of digital outreach intervention strategies (Aim 2) and the penetration, acceptability, and scalability of the digital outreach intervention strategies (Aim 3).

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Neil, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States